CLINICAL TRIAL: NCT02835209
Title: Effect of Position on the Spontaneous Breathing Trial
Brief Title: Positioning During SBT in NICU Infants
Status: Withdrawn | Type: Observational
Why Stopped: Change in clinical practice that logistically prevented this study from being engaged.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: DDD#603398
Record Dates: First submitted 2016-06-08; First posted 2016-07-18 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Distress Syndrome, Newborn; Ventilator-associated Lung Injury
Keywords: spontaneous breathing test; premature infant; work of breathing
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Work of breathing during SBT: Ventilated premature infants born 24 to 34+6 weeks gestational age.
  Interventions: Other: Work of breathing during SBT

INTERVENTIONS:
Other: Work of breathing during SBT — Pulmonary function tests and work of breathing indices will be collected during the spontaneous breathing test.

SUMMARY:
Mechanical ventilation is a life-sustaining intervention in premature infants with respiratory difficulties. There is relative consensus when to intubate and provide positive pressure mechanical ventilation in the presence of respiratory failure. In contrast, discontinuation of mechanical ventilation during recovery remains largely subjective. A potential predictive tool for neonatal extubation is the Spontaneous Breathing Trial (SBT). The efficacy of SBT or other tests used in older patient populations in improving clinical judgment is questionable in the neonatal population with its unique physiology, respiratory mechanics and drive factors. Christiana Care Health System NICU currently uses the SBT as a standard part of neonatal assessment for extubation from mechanical ventilation.

Infants in the CCHS NICU are routinely cared for in multiple positions (prone, supine, lateral) throughout the day. What is unknown is the impact of infant positioning on the SBT. An SBT performed in one position may not predict infant respiratory status after extubation in another position. Understanding the impact of infant positioning and work of breathing indices independently or in combination with an SBT will aid clinicians in decision-making and potentially decrease neonatal morbidity (inaccuracy with timing and safety of extubation). This pilot study will begin to explore these clinically relevant factors.

Objectives: This pilot study will investigate the (1) role of infant position on SBT score and (2) the relationship of work of breathing indices in reference to the SBT score and infant position.

DETAILED DESCRIPTION:
Mechanical ventilation is a life-sustaining intervention in premature infants with respiratory difficulties. There is relative consensus when to intubate and provide positive pressure mechanical ventilation in the presence of respiratory failure. In contrast, discontinuation of mechanical ventilation during recovery remains largely subjective. Typically 25% of infants weighing <1500g who are extubated using these criteria require reintubation suggesting that the ability of clinicians to predict successful extubation is limited. A potential predictive tool for neonatal extubation is the Spontaneous Breathing Trial (SBT). The efficacy of SBT or other tests used in older patient populations in improving clinical judgment is questionable in the neonatal population with its unique physiology, respiratory mechanics and drive factors.

Christiana Care Health System NICU currently uses the SBT as a standard part of neonatal assessment for extubation from mechanical ventilation.

The SBT used at CCHS is a non-invasive 5-minute test performed on an intubated infant. Respiratory rates (RR), expired tidal volume (Vte), heart rate, and oxygen saturation by pulse oximetry (SpO2) are recorded. An SBT is considered passed, when there is no apnea (defined as no respiratory effort for greater than 20 seconds), no bradycardia (defined as heart rate less than 100 for greater than 15 seconds), and the SpO2 has been maintained at greater than 85% or SBT VE greater than 60% than that of the mechanical VE.

Potentially confounding the SBT, and unstudied, is the effect of position (prone, supine, lateral). Similar to adults, infant position has a significant effect on the efficacy of spontaneous breathing. Infants in the CCHS NICU are routinely cared for in multiple positions (prone, supine, lateral) throughout the day. What is unknown is the impact of infant positioning on the SBT. An SBT performed in one position may not predict infant respiratory status after extubation in another position. Understanding the impact of infant positioning and work of breathing indices independently or in combination with an SBT will aid clinicians in decision-making and potentially decrease neonatal morbidity (inaccuracy with timing and safety of extubation). This pilot study will begin to explore these clinically relevant factors.

Work of breathing (WOB) indices can be non-invasively measured utilizing respiratory inductive plethysmography (RIP). WOB indices measured by RIP have been utilized by this research team for clinical and research purposes, including at CCHS. RIP entails that an infant breathe calmly while wearing soft elastic cloth bands that comfortably encircle the rib cage and abdomen. Contained within the bands is a flexible sinusoidal wire that measures motion. Measurements are taken for a minimum of 10 breaths, but preferable throughout the duration of the 5 minutes SBT.

Objectives: This pilot study will investigate the (1) role of infant position on SBT score and (2) the relationship of work of breathing indices in reference to the SBT score and infant position.

ELIGIBILITY:
Inclusion Criteria:

* Infants born 24+0 to 34+6 weeks gestation
* Intubated for a minimum of 24hrs
* Qualify for an SBT as standard of care.

Exclusion Criteria:

* Previous history of abdominal or chest surgery
* Congenital malformation of the chest or abdomen
* Neuromuscular disorder
* Current medications affecting neuro-muscular tone
* Unable to be positioned either prone, supine or lateral as determined by the attending neonatologist.

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants who are mechanically ventilated.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Impact of infant positioning on spontaneous breathing test (SBT) pass rates | Less than 1 hour
  SBT will be performed with the infant in 3 different positions (supine, prone, side-lying).
Impact of infant positioning on spontaneous breathing test (SBT) fail rates | Less than 1 hour
  SBT will be performed with the infant in 3 different positions (supine, prone, side-lying)

SECONDARY OUTCOMES:
WOB correlates of SBT pass rates | Less than 1 hour
  Pulmonary function tests will be performed during the SBT in each position (supine, prone and side-lying).
WOB correlates of SBT fail rates | Less than 1 hour
  Pulmonary function tests will be performed during the SBT in each position (supine, prone and side-lying).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Locke, DO, MPH, Principal Investigator — Christiana Care Health Services

IPD SHARING:
Plan to Share IPD: Yes
De-identified data would be shared in a data warehouse after a data use agreement was in place.